CLINICAL TRIAL: NCT01922401
Title: Effects of a Changes in Inspiratory to Expiratory Ratio on Respiratory Mechanics and Oxygenation During Laparosopic Bariatric Surgery
Brief Title: Inverse Ratio Ventilation on Bariatric Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, Assistant professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: GCIRB2013-164
Record Dates: First submitted 2013-08-08; First posted 2013-08-14 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- inverse ratio ventilation (Experimental): in one group change the I:E ratio during pneumoperitoneum 1:2-1:2-2:1
  Interventions: Other: inverse ratio ventilation

INTERVENTIONS:
Other: inverse ratio ventilation — change the I: E ratio 1:2-1:1-2:1

SUMMARY:
for evaluating inverse ratio ventilation of laparoscopic bariatric surgery

DETAILED DESCRIPTION:
inverse ratio ventilation had been improve the oxygenation and respiratory mechanics during care of ARDS patients or during general anesthesia. We hypothized inverse ratio ventilatio could improve the oxygenation and respiratory mechanics on the obese patient also.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS 1-2 obese patients(BMI>30)

Exclusion Criteria:

* underlying cardiopulmonary diasease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Arterial oxygenation (PaO2) | baseline PaO2-2hour after pneumoperitoneum
  sampling for arterial blood from arterial cannular weill be analysed 10 min after anesthetic induction, 20 min after pneurmoperitoneum (PP)with 1:2 of IE ratio, 20 min after after pneurmoperitoneum (PP)with 1:1 of IE ratio, after pneurmoperitoneum (PP)with 2:1 of IE ratio and end of operation

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Cheon Lee, M.D, Study Director — Gachon Universiy Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea